CLINICAL TRIAL: NCT05854134
Title: Effectiveness of Closed Chain Versus Aerobic Exercise for Strengthening and Improving Quality of Life in Post Stroke Patients
Brief Title: Effectiveness of CC VS Aerobic Exercise for Strengthening and Improving QOL in Post Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/533
Record Dates: First submitted 2023-03-18; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed Chain (Experimental)
  Interventions: Diagnostic Test: Closed Chain
- Aerobic Exercise (Other)
  Interventions: Diagnostic Test: Aerobic Exercise

INTERVENTIONS:
Diagnostic Test: Closed Chain — Effectiveness of Closed Chain for Strengthening and Improving Quality of Life in Post Stroke Patients
  Arms: Closed Chain
Diagnostic Test: Aerobic Exercise — Effectiveness of Aerobic Exercise for Strengthening and Improving Quality of Life in Post Stroke Patients
  Arms: Aerobic Exercise

SUMMARY:
To determine the effects of closed chain versus aerobic exercise for strengthening and improving quality of life in post stroke patients

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic post stroke patients (either left or right side)
* Patients of both gender
* Age range in between 40 to 60
* Patient with cognitive functioning

Exclusion Criteria:

* History of any cardiac problem
* Recurrent stroke
* Any kind of disability or amputated limb
* Neurological conditions like Parkinsonism, epilepsy and
* spinal cord injury.
* Any kind of fracture or dislocation history.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Barthel Index Scale | 6 Months
The Oxford Scale | 6 Months
  The Oxford Scale to improve QOL in Post Stroke Patients

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No